CLINICAL TRIAL: NCT04194775
Title: A Multi-Center, Double-Blind, Randomized, Phase III Study to Investigate the Efficacy and Safety of Nofazinlimab (CS1003) in Combination With Lenvatinib Compared to Placebo in Combination With Lenvatinib as First-Line Therapy in Subjects With Advanced Hepatocellular Carcinoma (HCC)
Brief Title: A Study of Nofazinlimab (CS1003) in Subjects With Advanced Hepatocellular Carcinoma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: CStone Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CS1003-305
Record Dates: First submitted 2019-12-10; First posted 2019-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — CS-1003

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nofazinlimab (CS1003) (Experimental)
  Interventions: Drug: Nofazinlimab (CS1003)+Lenvatinib
- Nofazinlimab (CS1003) placebo (Placebo Comparator)
  Interventions: Drug: Nofazinlimab (CS1003) Placebo+Lenvatinib

INTERVENTIONS:
Drug: Nofazinlimab (CS1003)+Lenvatinib — Nofazinlimab (CS1003), intravenous (i.v.) administration every 21 days; Lenvatinib oral administration, once daily
  Arms: Nofazinlimab (CS1003)
Drug: Nofazinlimab (CS1003) Placebo+Lenvatinib — Nofazinlimab (CS1003) Placebo, i.v. administration every 21 days ; Lenvatinib oral administration, once daily
  Arms: Nofazinlimab (CS1003) placebo

SUMMARY:
This is a multi-center, double-blind, randomized, phase III study to investigate the efficacy and safety of Nofazinlimab (CS1003) in combination with lenvatinib and placebo in combination with lenvatinib in the treatment of subjects with no prior systemic treatment and with unresectable advanced hepatocellular carcinoma (HCC). Subjects cannot be eligible for locoregional therapy. In this study, Nofazinlimab (CS1003) (or placebo) and lenvatinib are both considered as the study treatment while Nofazinlimab (CS1003) (or placebo) is the investigational product of and lenvatinib is selected as the basic treatment for HCC.

ELIGIBILITY:
Inclusion criteria

1. Age ≥18 years on the day of signing informed consent-(For Taiwan, the lower limit of age is 20 years).
2. Subjects with unresectable advanced HCC, that is not eligible for surgery and/or locoregional therapy (Stage B or C based on Barcelona Clinic Liver Cancer [BCLC] staging system, and meets either one of the following criteria: 1) histologically or cytologically confirmed diagnosis of HCC, 2) clinically confirmed diagnosis of HCC according to American Association for the Study of Liver Diseases (AASLD) criteria. Patients without cirrhosis require histological confirmation of diagnosis.
3. With at least one measurable lesion can be assessed
4. Eastern Cooperative Oncology Group performance status (ECOG PS) 0 or 1.
5. Life expectancy ≥ 3 months.
6. Child-Pugh A
7. No prior systemic treatment for advanced HCC
8. Subjects with hepatitis B virus (HBV) infection, are willing to continue receiving antiviral treatment while on study.
9. Subjects have adequate organ and marrow function. Female subjects with childbearing potential must have negative serum pregnancy test result at screening. Female subjects with childbearing potential, and male subjects and their female partners with childbearing potential must agree to use an contraceptive method(s) from the day of signing informed consent form (ICF), during the study and till at least 6 months after the last dose of study treatment.

   Exclusion criteria
10. Fibrolamellar-HCC, sarcomatoid, cholangiocellular carcinoma or mixed cholangiocarcinoma and HCC.
11. A prior bleeding event due to esophageal within 6 months or other gastrointestinal bleeding events within 28 days prior to screening.
12. Malabsorption syndrome or inability to take oral medication due to other causes.
13. HBV and HCV co-infection.
14. Investigator evaluates to increase the drug related risk caused by enrolling subjects in trial and taking study drug, or any serious or uncontrolled systematic disease that confound the drug absorption or the study outcome, e,g diabetes mellitus, hypertension, rheumatoid arthritis, major cardiovascular disease and so on.
15. Surgery or locoregional therapy for palliative purpose within 4 weeks prior to study treatment.
16. History of other malignancy(ies) in the past 5 years, except for malignant disease treated with curative intent and without active disease.
17. Known history of human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS).
18. Current or prior use of systemic corticosteroid (> 10 mg/day prednisone or equivalent) or other immunosuppressive medication within 14 days prior to the first dose of study treatment.
19. History of bone marrow transplantation or organ transplantation.
20. History of anaphylaxis or hypersensitivity to any ingredient of the investigational product.
21. Any contraindication of lenvatinib.
22. Known history of drugs abuse that would interfere with cooperation with the requirements of the trial.
23. Pregnant or lactating female subjects.
24. History of psychiatric disease that would interfere with cooperation with the requirements of the trial; lack of or with restricted physical capability.
25. QTc interval > 470 msec (as calculated with Fridericia's formula) at screening electrocardiogram (ECG);
26. Any condition that would in the investigator's judgment, prevent the subject from participating in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 534 (Actual)
Dates: Start 2019-12-13 (Actual); Primary Completion 2025-06-18 (Actual); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Expected to be 5.5 years after the first patient is enrollment.

SECONDARY OUTCOMES:
Objective response rate (ORR) assessed by blinded independent central review committee(BICR) | Expected to be 5.5 years after the first patient is enrollment.
Progression-free survival(PFS) assessed by blinded independent central review committee(BICR) based on Response Evaluation Criteria in Solid Tumors(RECIST) v1.1 | Expected to be 5.5 years after the first patient is enrollment.
Progression-free survival(PFS) evaluated by investigator based on RECIST v1.1 | Expected to be 5.5 years after the first patient is enrollment.
Objective response rate (ORR) evaluated by investigators based on RECIST v1.1 | Expected to be 5.5 years after the first patient is enrollment.
Duration of response (DoR) evaluated by blinded independent central review committee(BICR) based on Response Evaluation Criteria in Solid Tumors(RECIST) v1.1 | Expected to be 5.5 years after the first patient is enrollment.
Duration of response (DoR) evaluated by investigators based on Response Evaluation Criteria in Solid Tumors(RECIST) v1.1 | Expected to be 5.5 years after the first patient is enrollment.
Disease control rate (DCR) evaluated by blinded independent central review committee(BICR) based on Response Evaluation Criteria in Solid Tumors(RECIST) v1.1 | Expected to be 5.5 years after the first patient is enrollment.
Disease control rate (DCR) evaluated by investigators based on Response Evaluation Criteria in Solid Tumors(RECIST) v1.1 | Expected to be 5.5 years after the first patient is enrollment.
Percentage of Participants with Adverse Events | Expected to be 5.5 years after the first patient is enrollment.
Peak and trough serum concentrations of CS1003 | Expected to be 5.5 years after the first patient is enrollment.
Number and percentage of subjects who develop anti-CS1003 antibody (ADA) | Expected to be 5.5 years after the first patient is enrollment.
Time to deterioration (TTD), defined as the time from randomization to the first deterioration of European Organization for the Research and Treatment of Cancer (EORTC) Quality-of-Life Questionnaire Core 30 (QLQ-C30) scale | Expected to be 5.5 years after the first patient is enrollment.

CONTACTS AND LOCATIONS:
Locations (74):
- United States (5):
  - Southern California Research Center, Coronado, California
  - Inland Empire Liver Foundation, Rialto, California
  - Mercy Medical Center, Baltimore, Maryland
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - Stony Brook University Cancer Clinical Trials, Stony Brook, New York
- China (40):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - The First Affiliated Hospital Of Anhui Medical University, Hefei, Anhui
  - The Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Beijing You'an Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - The 900th Hospital of Joint Logistic Support Force of PLA, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Foshan First People's Hospital, Foshan, Guangdong
  - Nanfang Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou University of Traditional Chinese Medicine, Guangzhou, Guangdong
  - Guangxi Medical University Affiliated Tumor Hospital, Nanning, Guangxi
  - Hainan General Hospital - Hepatology, Haikou, Hainan
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Luoyang Central Hospital, Luoyang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Zhengzhou University - First Affiliated Hospital, Zhengzhou, Henan
  - hubei Cancer Hospital, Wuhan, Hubei
  - Tongji Hospital - Medical Oncology, Wuhan, Hubei
  - Hunan Cancer Hospital - Radiology, Changsha, Hunan
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - The First People's Hospital of Huai'an, Huai'an, Jiangsu
  - Nantong Tumor Hospital, Nantong, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Yanbian University Hospital, Yanbian, Jilin
  - Jinan Military Region General Hospital of the People's Liber, Jinan, Shandong
  - Shangdong Provicial Qianfoshan Hospital, Jinan, Shandong
  - Affiliated Hospital Of Jining Medical University, Jining, Shandong
  - Linyi Cancer Hospital, Linyi, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Cancer Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Eastern Hepatobiliary Surgery Hospital - Hepatology, Shanghai, Shanghai Municipality
  - Shanghai First People's Hospital, Shanghai, Shanghai Municipality
  - Sichuan University - West China Hospital, Chengdu, Sichuan
  - Tianjin Medical University - Cancer Institute & Hospital - Oncology, Tianjin, Tianjin Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
- Italy (5):
  - Azienda Unità Locale Socio Sanitaria n. 1 Dolomiti, Distretto di Feltre, Ospedale di Feltre, Feltre, Belluno
  - Istituto Oncologico Veneto IOV IRCCS - Medical Oncology Unit 1, Padua, Veneto
  - Casa di Cura Dott. Pederzoli S.p.A (Ospedale Pederzoli), Peschiera del Garda, Verona
  - PO di Cremona, ASST di Cremona - Oncologia - Cremona - Radiology, Cremona
  - Fondazione IRCCS Policlinico San Matteo, Pavia
- Poland (4):
  - MED-POLONIA Sp.z o.o., Poznan, Greater Poland Voivodeship
  - Centrum Badan Klinicznych, Wroclaw, Lower Silesian Voivodeship
  - Centrum Onkologii im. prof. F. Lukaszczyka, Bydgoszcz
  - Narodowy Instytut Onkologii im. Marii Skłodowskiej-Curie - Państwowy Instytut Badawczy, Warsaw
- Spain (14):
  - Complexo Hospitalario Universitario A Coruña, A Coruña, Galicia
  - Complejo Hospitalario Universitario de Orense, Ourense, Galicia
  - Hospital Universitario Puerta De Hierro De Majadahonda, Majadahonda, Madrid
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Ntra. Sra. de Sonsoles, Ávila
  - Hospital Del Mar, Barcelona
  - H.U. de Burgos, Burgos
  - ICO-Hospital Universitari de Girona Dr. Josep Trueta, Girona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario La Paz, Madrid
  - H.U.V.Arrixaca, Murcia
  - Hospital Universitario Virgen De La Macarena, Seville
  - Consorcio Hospital General Universitario de Valencia, Valencia
  - Hospital Unviersitario Miguel Servet, Zaragoza
- Taiwan (6):
  - China Medical University Hospital - Internal Medicine - Taichung, Taichung
  - Taichung Veterans General Hospital - Gastroenterology, Taichung
  - Chi Mei Hospital, Liouying - Department of Oncology, Tainan
  - Chi Mei Medical Center - YongKang - Gastroenterology - Gastroenterology, Tainan
  - National Cheng Kung University Hospital - Internal Medicine, Tainan
  - Tri-Service General Hospital - Neihu Branch - Pulmonary, Taipei